CLINICAL TRIAL: NCT03640611
Title: Investigating the Relation Between Environmental Factors and Activity-participation in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özge ÇANKAYA, Research assistant, Hacettepe University
Other Study IDs: Özge Çankaya
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy; Activity; Participation
Keywords: cerebral palsy, activity, participation, environmental factors, ICF-CY
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) is a chronic condition that causes the most childhood disabilities on worldwide. Impairment in movement and posture development seen in children with CP it causes difficulties in performing activities and affect in emotional, social, and cognitive abilities cause limited participation in everyday life. The ICF-CY child is divided into five categories: body structure and functions, activities, participation, environmental and personal factors, it is treated holistically. Initially, children with CP have adopted the view that environmental factors can also affect functionality, while focusing on the treatment of motor disorders to reduce activity and participation limitations in physiotherapy and rehabilitation applications. Environmental factors; the environment in which the child lives, his family, the devices he uses, health and care services, and government policies. These factors vary according to each country's own cultural and economic opportunities. The investigator planned to do this study because we found that there is a need for a comprehensive study of children with SP in Turkey, which does not reveal the relationship between environmental factors and activity and level of participation.

DETAILED DESCRIPTION:
The study consist of two phases:

1. European Child Environment Questionnaire (ECEQ) will translate in to Turkish in the first phase.

   * Forvard translation (translate to Turkish from English)
   * Expert opinion (Turkish version will control by expert)
   * Back translation (Turkish version will translate to English)
   * Cultural adaptation Validity and reliability study will done
2. The relationship between environmental factors and activity and participation will be investigated in the second phase.

Eligibility Criteria

* 2-18 years old
* Cerebral palsy diagnosed
* Children or family who understand and speek Turkish language
* Children or family who know writing and reading
* Volunteer to join the study

Outcome Measures

1. Clinical classifications:

   Gross Motor Function Classification System (GMFCS) for classifying gross motor function levels Manuel ability classification system (MACS) for classifying fine motor function levels Communication Function Classification System (CFCS) for classifying communication function levels Eating Drinking Abilities Classsification System (EDACS) for classifying eating and drinking functions levels will be used
2. Activity evaluation:

   Gross Motor Function Measurement (GMFM) Pediatric Evaluation of Disabilty Inventory (PEDI) will be used
3. Participation:

   Life Habits Questionnaire (Life-H) will be used
4. Environmental factors:

European Child Environment Questionnaire (ECEQ) Impact on Family Scale (IPFAM) will be used

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cerebral palsy
* Volunteer to join the study
* Know writing and reading
* speeking Turkish

Exclusion Criteria:

* Seconder neurologic impairment
* not complete the evaluation

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All types of cerebral palsy 20 children in each GMFCS levels
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
European Child Environment Questionnaire (ECEQ) | 20 minute
  60 item, created for evaluating environmental factors. Higher values means environmental factors aren't for child. The ECEQ total score changes between 0-120. There is no subscale in ECEQ.

CONTACTS AND LOCATIONS:
Overall Officials: ÖZGE ÇANKAYA, Principal Investigator — Hacettepe University
Locations (1):
- Özge Çankaya, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Cankaya O, Kerem Gunel M, Ozdemir P. Construct-concurrent validity and reliability of the European Child Environment Questionnaire (ECEQ) in a sample of Turkish children with cerebral palsy. Disabil Rehabil. 2022 May;44(10):2104-2112. doi: 10.1080/09638288.2020.1822930. Epub 2020 Sep 29. PMID 32988240